CLINICAL TRIAL: NCT02520583
Title: The Effects of Probiotic Supplementation on Markers of Muscle Damage and Performance Following Exercise Induced Muscle Damage
Acronym: PRO001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Jonathan Oliver, Assistant Professor, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 1509-009-1502
Record Dates: First submitted 2015-07-29; First posted 2015-08-13 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Probiotics
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- MICROBAC (Experimental): Bacterial cultures
  Interventions: Dietary Supplement: Lactic acid bacteria and bifidobacteria
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactic acid bacteria and bifidobacteria
  Arms: MICROBAC
Other: Placebo
  Arms: Placebo

SUMMARY:
To determine the effect of probiotic supplementation on the inflammatory response and subsequent performance following a muscle damaging exercise bout, a double-blind, randomized placebo controlled two-factor repeated measures design will be employed. The dependent variables for this study will include measures of performance as well as markers of inflammation in a single limb model. Participants who qualify for study participation will have their height, weight, and body composition assessed (skin fold) followed by baseline measurements for determination of isometric and dynamic strength. Initial limb will be determined randomly. Following baseline testing, participants will randomly be assigned to ingest either a probiotic or placebo. Supplementation will begin at least 24 hours post baseline testing. Twenty-one days after initiating supplementation, participants will again complete performance testing followed by an exercise bout known to elicit muscle damage and produce an inflammatory response. Participants will then repeat performance testing 24, 48, and 72 hours post muscle damaging bout. Blood samples for determination of markers of inflammation will be taken throughout study duration. Following a 3-week wash-out period (21 days), participants will repeat the experiment following the alternate supplement regimen with the contralateral limb.

DETAILED DESCRIPTION:
General Performance Testing and Muscle Damaging Exercise Bout Following familiarization and consenting procedures, participants will complete a series of performance tests designed to determine maximal performance. Those tests will include a test of isometric strength and dynamic strength of the elbow flexors. Isometric strength will be tested with subjects elbow at a fixed angle and measurement of the force the subject exerts, while dynamic strength with be a test of maximal strength through a specified range of motion. Prior to baseline testing, participants will be asked to refrain from any physical activity outside of daily living for the preceding 48 hours as well as eliminate products that contain caffeine and/or alcohol. These tests will be repeated over the course of the study as outlined in Table 1 to examine if supplementation with probiotics attenuates the loss in strength following the muscle damaging exercise bout. An exercise bout known to induce significant muscle damage (eccentric) of the elbow flexors will be performed on Day 22 of supplementation. This will be an eccentric based protocol in which the muscle is stretched while generating force to overcome the stretch. To avoid any carryover effect, the initial arm will be selected at random while the contralateral arm will be used during the crossover experimental trial.

Nutrition and Supplementation Following baseline performance measures, participants will be randomly assigned to ingest, in a double blind manner, either a probiotic supplement or placebo. Participants will begin supplementation 24 hours post baseline performance measures and will ingest the supplement (capsule form) once per day prior to consuming any food. Supplementation will continue for 25 days (21 days prior to post measures and 4 days of post testing). To ensure compliance, participants will report to the laboratory weekly and be provided individually wrapped supplement containers. Return of empty containers will be used to verify compliance. In addition, participants will complete a daily supplement adherence and adverse side effects questionnaire (Appendix) weekly upon reporting to the laboratory.

Blood Sampling and Inflammatory Markers A baseline blood sample will be obtained prior to any performance testing and supplementation. Further, on the day of the muscle damaging exercise bout, participants will provide a blood sample for baseline determination of inflammatory blood markers and muscle damage. Blood samples will also be taken immediately post, 30, and 60 minutes post damaging exercise bout. Participants will then return to the laboratory 24, 48, and 72 hours following exercise bout to provide additional blood samples. Thirty six milliliters will be sampled at each time blood is drawn. If an emergency were to arise, the laboratory protocol for emergency management will be followed.

Soreness and Swelling Assessment An algometer will assess deep muscle pain and trigger point tenderness of the biceps muscles resulting from muscle damage. The investigators will apply a pressure algometer at points on the muscle. The pressure threshold measurements will consist of the following steps. First, the following explanation will be given to each participant: 'I am going to measure pressure threshold; that is, how much pressure will induce discomfort. I am going to increase pressure slowly with this device. Say ''Yes'' when you start to feel pain or discomfort. I will stop the pressure as soon as you say ''Yes'', so it will not hurt you. It is important that you understand that this is a test of sensitivity, not a test of endurance. Do you understand or have any questions?' After the explanation is given, the algometer will be placed exactly over the indelible mark and perpendicular to the muscle under observation. Pressure will increase continuously at 1 kg per second until the participant says 'Yes'. At this time, the pressure will stop, the meter removed from the skin, and the measurement recorded. The mean of 1 measurement taken at each of the 3 sites will be recorded as the pressure pain threshold. The subjects will be blinded to their pressure pain measurements. Additionally, the resting angle of the arm will be measured along with arm circumference to determine degree of swelling.

ELIGIBILITY:
Inclusion Criteria:

* Participants must currently be participating in structured resistance training and must have been doing so for the previous 1 year period.

Exclusion Criteria:

* Having consumed any nutritional supplements and/or ergogenic aids for the preceding 6 week period.
* Having not taken any anti-inflammatory medications for the previous month.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Blood markers of muscle damage (cytokines, creatine kinase) | 1 year

SECONDARY OUTCOMES:
Isometric strength | 1 year
  Isometric strength will be assessed on a isokinetic dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian Universti, Fort Worth, Texas, United States

REFERENCES:
- [Derived] Jager R, Purpura M, Stone JD, Turner SM, Anzalone AJ, Eimerbrink MJ, Pane M, Amoruso A, Rowlands DS, Oliver JM. Probiotic Streptococcus thermophilus FP4 and Bifidobacterium breve BR03 Supplementation Attenuates Performance and Range-of-Motion Decrements Following Muscle Damaging Exercise. Nutrients. 2016 Oct 14;8(10):642. doi: 10.3390/nu8100642. PMID 27754427